CLINICAL TRIAL: NCT07015645
Title: Long-Term Outcomes of Hypopituitarism Following Gamma Knife Radiosurgery for Pituitary Adenomas
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Awad Mohamed Hegab, Lecturer of Neurosurgery, Faculty of Medicine, Al-Azhar University, Damietta, Egypt., Al-Azhar University
Other Study IDs: DFM-IRB 00012367-25-05-006
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Long Term; Hypopituitarism; Gamma Knife Radiosurgery; Pituitary Adenomas
MeSH Terms: conditions — Hypopituitarism; Pituitary Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pituitary Adenomas group: Patients received gamma knife radiosurgery (GKRS) treatment for pituitary adenomas.
  Interventions: Procedure: Gamma Knife Radiosurgery

INTERVENTIONS:
Procedure: Gamma Knife Radiosurgery — Patients received gamma knife radiosurgery (GKRS) treatment for pituitary adenomas.

SUMMARY:
This study aims to assess long-term outcomes of hypopituitarism following gamma knife radiosurgery (GKRS) for pituitary adenomas.

DETAILED DESCRIPTION:
Pituitary adenomas (PAs) are one of the most common intracranial neoplasms, accounting for 10-20% of diagnosed brain tumors.

Initial gamma knife radiosurgery (GKRS) can be an alternative treatment for selected NFPA patients with comorbidities, documented growth small tumors, cavernous sinus invasion, or advanced age.

Hypopituitarism is one of the most common complications of radiosurgery (Cordeiro et al., 2018). Long-term follow-up is crucial to assess new pituitary deficits. Typically, hypopituitarism presents within the first 2-4 years after the treatment with radiosurgery, but the risk of pituitary insufficiency increases to up to 80%. Reports on the highest incidence of new-onset hypopituitarism also mentioned the longest follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Both sexes.
* Patients treated with gamma knife radiosurgery (GKRS).

Exclusion Criteria:

* Patients with inadequate endocrine follow-up (<12 months).
* Patients who had undergone previous radiation therapy.
* Pituitary insufficiency which presents before gamma knife radiosurgery (GKRS).
* Patients without visible glands.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cohort study will be conducted in the Department of Neurosurgery, Al-Azhar University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of new-onset hypopituitarism | 5 years post-procedure
  Prevalence of new-onset hypopituitarism will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University (Damietta), Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.